## <u>Maternal Alcohol Reduction Intervention in</u> <u>South Africa [MaRISA]</u>



NCT05319977; May 18, 2021

Descriptive statistics will be used to describe the data for the overall sample and separately for participants enrolled while pregnant and postpartum. Data will be summarized using the mean (standard deviations) for continuous variables and percentages (frequency) for categorical variables. Changes from baseline to follow-up assessments on variables related to alcohol use and contextual/co-occurring issues (i.e., violence and depression) will be evaluated using the Cochran-Armitage Trend test. All analyses will be performed using SAS version 9.4.